CLINICAL TRIAL: NCT05692479
Title: Comparison of Physical Activity Self Worth of Women With and Without Premenstrual Syndrome
Brief Title: Premenstrual Syndrome and Physical Activity Self-Worth
Status: Completed | Type: Observational
Sponsor: Nigde Omer Halisdemir University (Other)
Collaborators: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Asli Celik, MSc. Lecturer, Nigde Omer Halisdemir University
Other Study IDs: 06.10.2022-14
Record Dates: First submitted 2023-01-11; First posted 2023-01-20 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Premenstrual Syndrome
Keywords: Premenstrual syndrome; women; self-worth; physical activity
MeSH Terms: conditions — Premenstrual Syndrome; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1 and Group 2: Women With and Without Premenstrual Syndrome
  Interventions: Other: Premenstrual Syndrome Scale, Women's Physical Activity Self-Worth Inventory, Descriptive data

INTERVENTIONS:
Other: Premenstrual Syndrome Scale, Women's Physical Activity Self-Worth Inventory, Descriptive data — Premenstrual Syndrome Scale, Women's Physical Activity Self-Worth Inventory, Descriptive data

SUMMARY:
Premenstrual syndrome (PMS) negatively affects the quality of life of millions of women. PMS is a common cyclic disorder characterized by somatic, cognitive, emotional and behavioral symptoms that usually occurs in young and middle-aged women, lasts during the luteal phase of the menstrual cycle and ends with the onset of menstruation.Studies have shown that women with high PMS symptoms are more inactive. Physical activity participation in women affects a wide spectrum of self-perceptions, including knowledge, social, and emotional self-perceptions. By determining which physical, emotional, social and academic/knowledge areas are affected by women, increasing their participation in physical activity can be achieved. The subject of the study is to determine the symptom severity of women with and without premenstrual syndrome and to examine how premenstrual syndrome affects physical activity self-worth.

DETAILED DESCRIPTION:
Premenstrual syndrome (PMS) negatively affects the quality of life of millions of women. PMS is a common cyclic disorder characterized by somatic, cognitive, emotional and behavioral symptoms that usually occurs in young and middle-aged women, lasts during the luteal phase of the menstrual cycle and ends with the onset of menstruation.Studies have shown that women with high PMS symptoms are more inactive. Physical activity participation in women affects a wide spectrum of self-perceptions, including knowledge, social, and emotional self-perceptions. By determining which physical, emotional, social and academic/knowledge areas are affected by women, increasing their participation in physical activity can be achieved. The subject of the study is to determine the symptom severity of women with and without premenstrual syndrome and to examine how premenstrual syndrome affects physical activity self-worth.

A total of 296 women age of 18-35 participate in the research. Participants were divide into two groups with and without premenstrual syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate in the study
* Being 18-35 years old
* Being women
* To be menstruating

Exclusion Criteria:

* Evaluation form missing
* Not menstruating for 12 months or more
* Having any psychological diagnosis
* Being pregnant

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Premenstrual syndrome occurs only in women.
Study Population: Premenstrual syndrome (PMS) negatively affects the quality of life of millions of women. PMS is a common cyclic disorder characterized by somatic, cognitive, emotional and behavioral symptoms that usually occurs in young and middle-aged women, lasts during the luteal phase of the menstrual cycle and ends with the onset of menstruation.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Descriptive Data | Baseline
  In the general evaluation form, data such as age, gender, weight, height, age at menarche, menstruation interval, menstrual pattern, presence of gynecological problems, presence of dysmenorrhea, pain level, exercise status, presence of chronic disease will be recorded.
Premenstrual Syndrome Scale | Baseline
  The Premenstrual Syndrome Scale (PMSS) was developed by Gençdoğan in 2006, based on DSM III and DSM-IV, and its validity and reliability were established. PMSS is a 44-item five-point Likert-type scale. After each item is read in PMSS, marking is made by taking into account the degrees to the right of the relevant item, depending on whether this situation is within the period of "one week before menstruation". In scoring the scale, "Never" is evaluated as 1, "Very little" as 2, "Sometimes" as 3, "Often" as 4, and "Constantly" as 5 points. A score of 138 or higher indicates PMS.
Women's Physical Activity Self-Worth Inventory | Baseline
  The Women's Physical Activity Self-Worth Inventory (Women's Physical Activity Self-Worth Inventory), developed by Huberty J. et al. in 2013, is a 37-item multidimensional scale. Turkish version study, validity and reliability were done by Yutçiçek and Kömürcü in 2019. FAESQ is a 37-item Likert-type (Strongly Disagree (1), Disagree (2), Agree, (3), Strongly Agree (4)) scale that evaluates the non-physical aspects of physical activity-related self-worth in women. The total score obtained from the scale varies between 37 and 148. As the score increases, the sense of self-worth increases.

CONTACTS AND LOCATIONS:
Overall Officials: Gürkan Demirtaş, MSc., Principal Investigator — Niğde Ömer Halisdemir University; Arife Akbulut, MSc., Principal Investigator — Ankara Yildirim Beyazıt University; Havva Sümeyye Eroğlu, MSc., Principal Investigator — Gazi University
Locations (1):
- Niğde Ömer Halisdemir University, Niğde, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No